CLINICAL TRIAL: NCT02301312
Title: A Clinical Investigation to Assess the Safety and Performance of POSS-PCU Small Diameter Grafts as Conduits in Arteriovenous (AV) Access
Brief Title: Clinical Study of POSS-PCU Vascular Grafts for Vascular Access
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14/0276
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2019-10

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POSS-PCU graft (Experimental): POSS-PCU vascular graft will be used to create vascular access for dialysis.
  Interventions: Device: POSS-PCU vascular graft

INTERVENTIONS:
Device: POSS-PCU vascular graft — New vascular access graft

SUMMARY:
This study evaluates the safety and performance of a new vascular graft made of POSS-PCU as a vascular access conduit for haemodialysis. 30 patients requiring access for dialysis will be enrolled and monitored at regular intervals for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects requiring vascular access for haemodialysis
* Subjects with no suitable vein.
* Subjects aged 18 - 80 years old
* Subjects are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained
* Patients of child bearing potential, who are sexually active, must agree to the use of 2 highly effective forms of contraception throughout their participation in the study and for 6 months after completion of treatment:

  * Condom with spermicide.

AND 1 of the following:

* Oral contraceptive or hormonal therapy (e.g. hormone implants).
* Placement of an intra-uterine device.

Exclusion Criteria:

* Subjects with predicted short-term survival (less than 18 months) or poor prognosis (this will be on the discretion of the clinician in charge)
* Subjects with left ventricle ejection fraction (LVEF) <20% diagnosed on ECHO either pre-procedure or documented within the previous 3 months prior to consent.
* Pregnant or lactating
* Allergies to any constituents of the graft material
* Patients who are infected or colonized with Methicillin Resistant Staphylococcus Aureus (MRSA).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Patency rate | 18 months
  The primary performance end point of the study is the patency rate of the POSS-PCU graft at the end of the 18 months as measured with US Doppler, which will be compared to the known patency rate for the PTFE graft
Safety endpoint of this study is defined as any Serious Adverse Event related to the implantation procedure or device implantation within 30 days of implantation procedure | 30 days

SECONDARY OUTCOMES:
Patency rate | 12 months
  Patency rate of POSS-PCU Graft at 2weeks, 3, 6, and 12 months as measured with US Doppler.
Secondary patency rate | 18 months
  Any surgical or endovascular intervention required to maintain the patency of the grafts up to the 18 month time point.

REFERENCES:
- [Derived] Askari F, Shafieian M, Solouk A, Hashemi A. A comparison of the material properties of natural and synthetic vascular walls. J Mech Behav Biomed Mater. 2017 Jul;71:209-215. doi: 10.1016/j.jmbbm.2017.03.016. Epub 2017 Mar 23. PMID 28347955